CLINICAL TRIAL: NCT04253106
Title: Liquid Biopsies (blood, Gastric Fluid) for the Personalized Management of Patients with Hereditary Diffuse Gastric Cancer: a Pilot Project
Brief Title: Liquid Biopsies for the Personalized Management of Patients with Hereditary Diffuse Gastric Cancer
Acronym: LISA-HDGC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: APHP190483
Record Dates: First submitted 2020-01-31; First posted 2020-02-05 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Hereditary Diffuse Gastric Cancer
Keywords: gastrectomy; somatic mutations; endoscopy; biopsies; methylation profil
MeSH Terms: conditions — Stomach Neoplasms | interventions — Liquid Biopsy; Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: Multicentric, prospective non-randomized study prognostic aim. Control group planned to have standard values.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Unaffected carriers of constitutional mutations (Experimental): Patients with CDH1 or CTNNA1 germline pathogenic variant. No history of diffuse gastric cancer.
  Interventions: Genetic: Liquid biopsies (blood, gastric fluid).
- All patients with FOGD (Active Comparator): without observation of macroscopic lesions paired with cases (age and sex)
  Interventions: Genetic: Liquid biopsies (blood, gastric fluid).

INTERVENTIONS:
Genetic: Liquid biopsies (blood, gastric fluid). — Next generation sequencing of a panel of diffuse gastric cancer genes, methylation analysis. Samples collected during routine screening endoscopy.

SUMMARY:
Activating somatic mutations and methylation profiles identified by liquid biopsies could identify CDH1 and CTNNA1 pathogenic variants carriers with invasive diffuse gastric cancer undetectable by upper G-I endoscopy.

DETAILED DESCRIPTION:
Carriers of germline pathogenic variants in the CDH1 and CTNNA1 genes have the Hereditary Diffuse Gastric Cancer Syndrome. Asymptomatic carriers have at high lifetime risk of diffuse gastric cancer (30-70%). Screening upper gastrointestinal endoscopy, even with multiple random biopsies, misses signet ring cell cancer foci. Invasive cancers can thus go undetected. There is therefore a recommendation of total risk-reducing gastrectomy, at least in carriers with a family history of gastric cancer. Novel screening strategies are needed. In this pilot project, the investigators will perform liquid biopsies of both blood and gastric fluid in asymptomatic carriers who refuse gastrectomy and in controls. The investigators aim to show that somatic mutations in a panel of genes involved in gastric cancer and methylation profiles are detected in a subset of carriers, and not in controls. These could be indicative of invasive cancer undetected by endoscopy, and would thus be a strong argument for risk-reducing gastrectomy. On the contrary, in the absence of somatic mutations in liquid biopsies, endoscopic surveillance could continue.

ELIGIBILITY:
Inclusion Criteria:

Case:

* Patient ≥ 18 years old
* CDH1 or CTNNA1 germline pathogenic variant.
* No history of diffuse gastric cancer.
* French social security.
* Ability to understand and willingness to sign a written informed consent document.

Volunteers:

* Patients ≥ 18 years old
* Patients with no oncological history
* Patients with macroscopically normal oeso-gastroduodenal fibroscopy
* French social security.
* Ability to understand and willingness to sign a written informed consent

Exclusion Criteria: for both arms

* Patients with cancer being treated
* Patients with metastatic cancer
* Medical contraindication to general anesthesia or FOGD (bleeding disorder, pregnant women )
* Patients under guardianship or curator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2020-11-26 (Actual); Primary Completion 2024-04-10 (Actual); Study Completion 2024-04-10 (Actual)

PRIMARY OUTCOMES:
Number of subjects in whom somatic mutations or methylation profiles are detected. | Over two years of surveillance

SECONDARY OUTCOMES:
Replicability of observations over successive endoscopies. Correlation between blood and gastric fluid. | Over two years of surveillance

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital Pitié Salpetrière, Paris, Paris, France

IPD SHARING:
Plan to Share IPD: Yes
The procedures carried out with the French data privacy authority (CNIL, Commission nationale de l'informatique et des libertés) do not provide for the transmission of the database, nor do the information and consent documents signed by the patients.
  Consultation by the editorial board or interested researchers of individual participant data that underlie the results reported in the article after deidentification may nevertheless be considered, subject to prior determination of the terms and conditions of such consultation and in respect for compliance with the applicable regulations.
Supporting Information: Study Protocol, ICF
Time Frame: Beginning 3 months and ending 3 years following article publication. Requests out of these time frame can also be submitted to the sponsor.
Access Criteria: Researchers who provide a methodologically sound proposal.